CLINICAL TRIAL: NCT01734681
Title: An Open-Label, Single-Arm, Phase 2 Study of G-202 in Patients With Chemotherapy-Naïve Metastatic Castrate-Resistant Prostate Cancer
Brief Title: Phase 2 Study of G-202 in Patients With Chemotherapy-Naïve Metastatic Castrate-Resistant Prostate Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: GenSpera, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: G202-002
Record Dates: First submitted 2012-11-19; First posted 2012-11-28 (Estimated); Last update posted 2014-02-19 (Estimated); Status verified 2013-02

CONDITIONS: Prostate Cancer.
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment with G-202 (Experimental): G-202 will be administered by intravenous infusion over one hour on Days 1, 2 and 3 of a 28-day treatment cycle. The G-202 dose will be 40 mg/m2 on Day 1 and 66.8 mg/m2 on Days 2 and 3.
  Interventions: Drug: G-202

INTERVENTIONS:
Drug: G-202

SUMMARY:
Prostate cancer that has returned after local treatment usually responds to hormone blocking treatment, but most patients eventually experience disease progression. Further chemotherapy does not normally lead to a cure or dramatic improvement in the disease and there is a need to identify new drugs that are beneficial for these patients without unacceptable side effects. Prodrug chemotherapy is an approach in which an inactive non-toxic agent is administered to the patient and gets activated within the body at specific locations, resulting in a higher concentration of the cytotoxic form at a tumour location whilst avoiding general side effects. G-202 is an example of prodrug chemotherapy. It does not have many general side effects because it is converted to a cell toxin only at the tumour or other specific locations in the body. G-202 is activated by Prostate Specific Memory Antigen (PSMA), a substance expressed by prostate cancer cells and in the blood vessels of most solid tumours, but not by normal cells or blood vessels in normal tissue. It is believed that activation of the prodrug G-202 will allow the drug to kill cancer cells, particularly prostate cancer cells. This study will evaluate the activity and safety of G-202 in men with castration-resistant prostate cancer (CRPC), which means the cancer has progressed after hormone blocking treatment, but who have not yet received chemotherapy and who have no or only a few symptoms from their CRPC. The study will evaluate clinical activity and safety of G-202 administered on three consecutive days of a 28-day cycle.

DETAILED DESCRIPTION:
Patients will undergo a screening period of up to 4 weeks. Patients who are deemed eligible will be entered into the study and undergo treatment with G-202. G-202 will be administered by intravenous infusion over one hour on Days 1, 2 and 3 of a 28-day treatment cycle. The G-202 dose will be 40 mg/m2 on Day 1 and 66.8 mg/m2 on Days 2 and 3.

The primary objective of the study is to determine the percentage of patients with chemotherapy-naïve metastatic castrate-resistant prostate cancer who do not have disease progression (radiographic or clinical) after 24 weeks of treatment with G-202.

A two-stage study design will be used to evaluate the percentage of patients who do not have disease progression after 24 weeks of treatment with G-202. If the percent of patients who are progression-free at 24 weeks is at most 15%, then the clinical efficacy of G-202 in this patient population will be considered unacceptably low. If, on the other hand, the percent of patients who are progression-free at 24 weeks is at least 35%, this will be considered sufficient evidence to consider further clinical investigation. The null hypothesis that the percent of patients who are progression-free at 24 weeks is at most 15% will be tested against the alternative hypothesis that the percent is greater than 15% at the one-sided 10% significance level. In order to avoid a suspension in accrual awaiting interim analysis, a two-stage study design for evaluating survival probabilities with continual accrual will be used.

An interim analysis for futility will be conducted after 24 evaluable patients have been accrued assuming that the time between accrual of the first patient and accrual of the 24th patient is at least 8 months. If 24 patients are accrued in less than 8 months, accrual will continue until the time period between the date of accrual of the first patient and the date of accrual of the last patient is at least 8 months. If the trial is not terminated for futility after the interim analysis, an additional 10 patients will be accrued for a total of 34 patients. The two-stage design minimizes the expected duration of accrual under the null hypothesis.

For the interim analysis, any patient who discontinues participation for reasons other than safety or disease progression before completing three full cycles and undergoing the 12-week follow-up assessment will be replaced. Any replaced patient will be included in all study analyses of the intent-to-treat and safety populations.

Safety will be assessed by the reporting of adverse events, vital signs and assessment of findings on physical exam and routine laboratory determinations. The severity of adverse events and laboratory findings will be assessed according to NCI Common Toxicity Criteria for Adverse Effects (CTCAE) V4.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed prostate adenocarcinoma
* Asymptomatic or minimally symptomatic
* Radiographic metastatic or recurrent disease
* Chemically- or surgically-castrated with disease progression
* Castrate testosterone level <50 ng/dL
* Discontinued flutamide, bicalutamide and nilutamide
* Absence of known brain metastases
* Age ≥18 years
* Eastern Cooperative Oncology Group performance status ≤ 2
* Estimated life expectancy ≥ 6 months
* Adequate hematopoietic function as demonstrated by:

  * hemoglobin of ≥ 9.0 g/dL without need for sustained blood transfusions
  * platelet count ≥100,000 platelet/mm3 (100 x 109/L)
  * White Blood Cell (WBC) count ≥ 2.0 x109/L and Absolute Neutrophil Count (ANC) ≥1.5 x109/L
* Adequate hepatobiliary function as demonstrated by:

  * Total bilirubin level ≤1.5 times the upper limit of normal (ULN), unless the patient has Gilbert's syndrome in which case the patient must have a total bilirubin level ≤ 2.5 x ULN
  * alanine aminotransferase (ALT) levels ≤ 2.5 x ULN
* Adequate renal function as demonstrated by creatinine level ≤1.5 x ULN or creatinine clearance (measured or calculated by Cockcroft-Gault formula) ≥ 50mL/min
* Acceptable coagulation profile (PT or INR, PTT < 1.5 x ULN)
* If of reproductive capacity, willing to use an effective double barrier method of birth control (i.e., latex condom, diaphragm, cervical cap, etc) during the study and for 30 days after the last administration of G-202

Exclusion Criteria:

* Prior chemotherapy
* Other concurrent therapy for prostate cancer other than LHRH agonists or antagonists.
* Treatment with therapeutic radionucleotides within 12 weeks of study entry
* Radiation therapy < 4 weeks before study entry
* Documentation of keratosis follicularis
* Pre-existing cardiac condition:
* use of inhibitors or inducers of cytochrome (CYP3A4) iso-enzymes
* Chronic use of opioids for cancer-related pain
* Corrected QT interval > 470 msec
* Active uncontrolled infection, including known history of AIDS, hepatitis B or C
* Proteinuria level > +2 on urine analysis

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-05; Primary Completion 2015-01 (Estimated); Study Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients who are progression-free after 24 weeks of treatment with G-202 | 24 weeks
  Determine the percentage of patients with chemotherapy-naïve metastatic castrate-resistant prostate cancer who do not have disease progression (radiographic or clinical) after 24 weeks of treatment with G-202

SECONDARY OUTCOMES:
Maximum prostatic specific antigen (PSA) change from baseline at any time | Every 4 weeks
Percent change in PSA from baseline to 24 weeks | 24 weeks
Time to PSA progression | Every 4 weeks
PSA Doubling time | Every 4 weeks
Best Objective Response | Every 12 weeks
Time to Disease Progression | Every 12 weeks
Progression Free Survival | Every 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Texas Health Science Center, San Antonio, Texas, United States